CLINICAL TRIAL: NCT06342531
Title: More Effective Violence Risk Management for Psychiatric Wards - eDASA+APP FI
Brief Title: More Effective Violence Risk Management - eDASA+APP FI
Acronym: eDASA+APP FI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tella Lantta, Adjunct Professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 210324
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Violence
Keywords: violence risk assessment; DASA; Dynamic Appraisal of Situational Aggression; mental health nursing; EPIC; electronic health records; violence risk management; inpatient psychiatric care; coercive measures; clinical decision support system; CDSS; co-design; nurse-patient collaboration

STUDY DESIGN:
Intervention Model Description: A pre-post design (quasi-experimental), a cluster design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- eDASA+APP FI (Experimental): Nurses in the study wards are using a CDSS 'eDASA+APP FI' in their daily clinical work to aid their short-term violence risk assessment and management, together with a patient if possible, to identify patients at elevated risk for violence in the coming 24 hours and to decrease (or maintain low) the risk with evidence-based, non-invasive nursing interventions.
  Interventions: Behavioral: eDASA+APP FI

INTERVENTIONS:
Behavioral: eDASA+APP FI — A CDSS for nurses to assist in their daily short-term violence risk assessment and management, is integrated into an EPIC-based EHR system.

SUMMARY:
The main goal of this study is to evaluate if the Finnish version of eDASA+APP (electronic Dynamic Appraisal of Situational Aggression + Aggression Prevention Protocol), a clinical decision support system (CDSS), has an impact on reducing workplace violence, use of coercive measures and increasing nurses' job satisfaction in adult psychiatric inpatient care.

DETAILED DESCRIPTION:
The study includes three phases: 1) exploring attitudes of nurses and nurse managers towards validated tools, violence risk assessment and management, 2) a pre-implementation including a co-design process of the eDASA+APP to ensure optimal integration and adaptation to local context and integration into the local EPIC based EHR system together with relevant stakeholders (health care staff and expert-by-experience), and 3) a quasi-experimental implementation study to evaluate the impact of the intervention (eDASA+APP FI).

ELIGIBILITY:
Inclusion Criteria:

* adult psychiatric wards

Exclusion Criteria:

* psychiatric wards specialized only for the care of people with intellectual disabilities, wards providing care for both adults and underaged patients (eating disorder units)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Workplace violence | Pre-post (3 months)
  Violence experienced by healthcare staff in the wards, routinely collected data

SECONDARY OUTCOMES:
Coercive measures | Pre-post (3 months)
  Routinely monitored and collected by the wards according to the Finnish Mental Health Act
Job satisfaction | Pre-post (3 months)
  Nurses yearly job satisfaction survey will be used (Nurse Engagement Survey (NESplus))

CONTACTS AND LOCATIONS:
Overall Officials: Tella Lantta, PhD, Principal Investigator — Department of Nursing Science, University of Turku, Finland
Locations (1):
- HUS University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffith JJ, Meyer D, Maguire T, Ogloff JRP, Daffern M. A Clinical Decision Support System to Prevent Aggression and Reduce Restrictive Practices in a Forensic Mental Health Service. Psychiatr Serv. 2021 Aug 1;72(8):885-890. doi: 10.1176/appi.ps.202000315. Epub 2021 May 17. PMID 33993715